CLINICAL TRIAL: NCT00034489
Title: A Phase II Study of a Combination of MTA (LY231514) and Gemcitabine in Patients With Metastatic Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2245; H3E-MC-JMCF
Record Dates: First submitted 2002-04-29; First posted 2002-04-30 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Breast Neoplasms
Keywords: metastatic breast cancer; combination therapy; Alimta
MeSH Terms: conditions — Breast Neoplasms | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: pemetrexed
Drug: gemcitabine

SUMMARY:
This is a study to explore how well the combination of LY231514 and Gemcitabine work together in patients with breast cancer that has spread beyond the location of the original tumor. Patients must have previously received treatment with anthracycline and taxane chemotherapy drugs.

DETAILED DESCRIPTION:
Gemcitabine is given by vein over 30 minutes on days 1 & 8 of each 21-day cycle. LY231514 is also given by vein over 10 minutes on day 8, following the Gemcitabine injection. Vitamin supplementation with oral folic acid and injectable B12 is initiated 7-10 days prior to the first dose of LY231514, and continuing throughout the patient's participation. Vitamin B12 is administered approximately every 9 weeks after the first injection. Appropriate antiemetic medication should be given to all patients. Dexamethasone 4mg PO twice daily is given for 3 days per cycle, beginning 1 day prior to LY231514 dosing. This is given to prevent or lessen the possibility of a rash.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of breast cancer
* measurable disease
* received prior anthracycline and taxane
* life expectancy > 3 months
* acceptable lab results

Exclusion Criteria:

* >3 prior regimens
* prior treatment with protocol drugs
* prior (pelvic) radiation
* active CNS metastasis
* inability to take oral vitamins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester, Minnesota, United States